CLINICAL TRIAL: NCT01949376
Title: Hippocampal Predictors of Cognitive Impairment (HippoPCI) in Breast Cancer Patients
Brief Title: Mild Cognitive Impairment in Breast Cancer Patients
Acronym: HippoPCI
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Lei Wang, Associate Professor, Northwestern University
Other Study IDs: 1R01NR014182-01 (NIH); 1R01NR014182-01 (NIH)
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer; Cognitive Impairment
Keywords: breast cancer; invasive ductal carcinoma; cognitive impairment; adjuvant therapy; hormone therapy; hormonal therapy; chemotherapy; chemo brain; MRI
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- HT Patients: any stage of breast cancer without brain metastasis, will undergo hormonal therapy without chemotherapy
- CT and HT Patients: any stage of breast cancer without brain metastasis, will undergo chemotherapy and hormonal therapy
- CT Patients: any stage of breast cancer without brain metastasis, has undergone surgery prior to screening, will undergo chemotherapy without hormonal therapy
- RT or NT Patients: any stage of breast cancer without brain metastasis, will not undergo chemotherapy or hormonal therapy; may undergo radiation therapy or have no therapy
- Controls: healthy, cognitively normal subjects

SUMMARY:
The purpose of this study is to improve our understanding of potential changes in size, shape and activity in some brain areas that can occur in women receiving different types of Breast Cancer therapy, and how these changes are related to the development of mild cognitive impairment as the result of these treatments.

DETAILED DESCRIPTION:
This study aims to identify neuroimaging biomarkers for predicting mild cognitive impairment (MCI) in breast cancer patients receiving adjuvant chemo and/or hormonal therapy by examining hippocampal-cortical neurocircuitry. Adjuvant therapies increase long-term survival, but produce changes in cognitive function in 30% (up to 70%) of women on average with breast cancer. Cognitive decline negatively impacts quality of life in patients and their supporters. Therefore, early identification of patients at risk for developing treatment-related cognitive impairment is needed to develop potential prevention or treatment options and prevent further decline. Our recent work demonstrates that patients receiving adjuvant hormonal treatment exhibit decline in cognition as soon as three months post treatment. Although neuroimaging studies have identified brain changes associated with chemotherapy ("chemo brain", no investigation has assessed the type and severity of such changes following hormonal therapy, nor has any study determined which individuals are at greatest risk for cognitive impairment.

Our central hypothesis is that measures of the hippocampal-cortical integrity can be used to predict cognitive decline, and changes of specific domains of cognitive performance in patients receiving adjuvant therapy over time will be related to changes in specific components of this circuitry over time.

ELIGIBILITY:
Inclusion Criteria:

* Female, within the age range of 40-70
* HT Patients - any stage of breast cancer without brain metastasis, will undergo hormonal therapy without chemotherapy
* CT and HT Patients - any stage of breast cancer without brain metastasis, will undergo chemotherapy and hormonal therapy
* CT Patients - any stage of breast cancer without brain metastasis, has undergone surgery prior to screening, will undergo chemotherapy without hormonal therapy
* RT or NT Patients - any stage of breast cancer without brain metastasis, will not undergo chemotherapy or hormonal therapy; may undergo radiation therapy or have no therapy
* Controls - cognitively normal on the basis of annual neuropsychological and research neurological examinations done as part of the Uniform Data Set (UDS), of the NIA Alzheimer's Disease Centers (ADC) program, recruited from the NU CNADC Clinical Core.
* All subjects must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

* Individuals who report significant medical, neurologic, or psychiatric illness, including but not limited to:
* Major depression
* Schizophrenia
* ADHD
* Autism
* Alzheimer's disease
* Dementia
* Obsessive-compulsive disorder
* Post-traumatic stress disorder
* Individuals with an Inventory of Depressive Symptomatology - Self Report (IDS-SR) score of 30 or higher, since this level of depression could affect cognitive test performance.
* Brain surgery or head injury

  * Individuals reporting previous head injury
  * Individuals requiring neurosurgical procedures
* Ineligibility for MRI scanning, including but not limited to:

  * Individuals who have non-MRI compatible medical implants or devices
  * Individuals who have any potential metal in their bodies
  * Individuals who have claustrophobia
  * Individuals with permanent makeup
* Individuals reporting consumption of drugs that would affect cognition (neuropsychiatric or illicit)
* Individuals indicating a history of breast cancer will be excluded from the healthy control group
* Women who are pregnant or are planning to become pregnant during study.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the following sites, all affiliated with Northwestern University Feinberg School of Medicine (NUFSM): a) outpatient facility at Galter Pavilion of Northwestern Medicine; b) Maggie Daley Center for Women's Cancer Care at Prentice Women's Hospital; and c) Lynn Sage Comprehensive Breast Cancer Center at Prentice Women's Hospital.
  Participants will also be recruited a) via advertisement in local newspapers, craigslist, Robert H. Lurie Comprehensive Cancer Center (RHLCC) Cancer Survivorship Institute website, and at community programs that serve cancer patients, including hospitals and support groups; and b) from community educational events sponsored by RHLCC, Women's Health Research Institute, and Cognitive Neurology and Alzheimer's Disease Center (CNADC).
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2013-06; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rates of change in cognitive function from before treatment to after treatment initiation | approximately 6 months
  Measured using a neuropsychological test battery

SECONDARY OUTCOMES:
Rates of change of brain structure from before treatment to after treatment initiation | approximately 6 months
  Measured using structural MRI scan
Rates of change of brain function from before treatment to after treatment initiation | approximately 6 months
  Measured using a functional MRI scan

CONTACTS AND LOCATIONS:
Overall Officials: Lei Wang, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No